CLINICAL TRIAL: NCT06200246
Title: Cardio-vascular Energy Transfer and Ventriculo-arterial Coupling in Heart Failure
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Other Study IDs: 480738
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure, Left-sided
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this pilot study is to investigate energy transfer fram the ventricle to the arteries in patients with heart failure, primary by investigating the total power.

ELIGIBILITY:
Inclusion Criteria:

Acute left ventricular failure due to:

* Myocardial ischemia
* Cardiomyopathy
* Myocarditis Sinus rhythm Age >18 years

Exclusion Criteria:

Cardiogenic shock Mechanical circulatory support Respiratory treatment Inotropic infusions Tachyarrhythmias Lack of capacity to consent

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises individuals experiencing decompensated heart failure within the first three days of hospital admission. It includes both newly diagnosed cases and individuals with a pre-existing heart failure diagnosis. The population is diverse, both regarding gender and etiology.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Cardio vascular energy transfer in heart failure patients. | During first 1-3 days after admission to hospital because of decompensated heart failure.
  We are investigating cardio vascular energy transfer in heart failure patients by calculating total power.

CONTACTS AND LOCATIONS:
Locations (1):
- St Olav hospital, Trondheim, Norway